CLINICAL TRIAL: NCT06489925
Title: Cerebrolysin as an Add-On Therapy to Standard Treatment of Posterior Circulation Stroke Secondary to Basilar Artery Occlusion
Brief Title: Cerebrolysin as an Add-On Therapy to Standard Treatment of Basilar Artery Occlusion
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Collaborators: Ever Neuro Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Marina Roje Bedekovic, Professor Marina Roje Bedeković, MD, PhD, neurologist, University Hospital Sestre Milosrdnice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 251-29-11/3-24-08
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Basilar Artery Occlusion; Posterior Circulation Brain Infarction
Keywords: Cerebrolysin; neuroprotection; basilar artery occlusion; add-on therapy; posterior circulation stroke
MeSH Terms: conditions — Brain Infarction | interventions — cerebrolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebrolysin group (Experimental): Patients with acute basilar artery occlusion who meet the eligibility criteria will receive Cerebrolysin in a single-day dosage of 30 ml, diluted with 250 ml of 0.9% saline intravenously in the first 24 hours after the stroke. Cerebrolysin will be further administered in the same dosage once daily in the morning for 14 consecutive days.
  Interventions: Drug: Cerebrolysin

INTERVENTIONS:
Drug: Cerebrolysin — The Cerebrolysin will be administered at least one hour after the standard treatment and no later than 24 hours after the stroke symptom onset.
  Other Names: Cerebrolysin®

SUMMARY:
The standard therapy for acute ischemic posterior circulation stroke (PCS) often leads to poor functional outcomes and high mortality rates, despite all advances in reperfusion therapy. Recent trials have shown that adding Cerebrolysin, a cerebral neuroprotective agent, to standard therapy for patients with acute ischemic anterior circulation stroke is safe and leads to improved functional outcomes. The purpose of this study is to assess the effectiveness and safety of Cerebrolysin with standard treatment for patients with PCS secondary to basilar artery occlusion (BAO).

The plan is to conduct a prospective, single-center, single-arm, open-label study with 20 acute basilar artery occlusion patients and premorbid modified Rankin Score (mRS) ≤3, treated with standard treatment (mechanical thrombectomy ± intravenous alteplase or conservative treatment) and Cerebrolysin as add-on therapy, compared with historical controls. Besides standard acute stroke assessment, standard treatment, and rehabilitation, the participants who meet the eligibility criteria will receive Cerebrolysin in a single-day dosage of 30 ml intravenously for 14 consecutive days. The participants will be closely monitored, and neuroimaging findings and clinical outcomes will be obtained during the drug administration period, on discharge, one month, and 3 months after the treatment onset.

The primary endpoints are mRS (0-3) on day 90 and mortality rate 90 days after the stroke onset. The secondary endpoints are defined as a change in any type of intracerebral bleeding and a change of min. 2 points on the National Institutes of Health Stroke Scale 24 hours, 14 days, 30 days, and 90 days post-stroke.

The investigators hypothesize that adding Cerebrolysin to standard stroke treatment will improve clinical outcomes and reduce morbidity and mortality in patients with acute basilar occlusion compared to standard treatment alone.

DETAILED DESCRIPTION:
The investigators plan to conduct a prospective, single-center, single-arm, open-label study with 20 acute basilar artery occlusion patients with premorbid modified Rankin Score (mRS) ≤3, treated with standard treatment (mechanical thrombectomy ± intravenous thrombolysis with alteplase or conservative treatment) and Cerebrolysin as add-on therapy, compared with historical controls.

All participants will receive the same standard of care and will be treated according to the latest European Stroke Organisation and American Stroke Organisation guidelines on acute stroke.

Besides standard acute stroke assessment, treatment, and acute rehabilitation, the participants who meet the eligibility criteria, are informed about the study and its potential risks, and have written informed consent, will receive Cerebrolysin in a single-day dosage of 30 ml intravenously for 14 consecutive days. The Cerebrolysin administration will start no earlier than one hour after the standard treatment, and no later than 24 hours after the stroke symptom onset. All possible side-effects will be closely monitored and in case of any adverse effect, the drug administration will be stopped, and the participant will be excluded from the further trial.

The participants will be closely monitored and the data on possible drug side effects, adverse effects, clinical findings, laboratory findings, and neuroimaging findings will be stored in the centralized hospital database. The clinical assessment and imaging analysis will be performed by an unbiased third-party neurologist/neuroradiologist.

The clinical findings and outcomes will be quantified by the National Institutes of Health Stroke Scale (NIHSS) 24 hours, 14 days, 30 days, and 90 days post-stroke and by the Modified Rankin Scale on discharge and 90 days post-stroke. The participants will undergo CT/ MRI neuroimaging for intracranial bleeding detection during admission, 24 hours after the stroke, and on discharge from the hospital. An additional imaging will be performed if indicated.

The interventional group and historical controls will be matched 1:1 based on the site of the basilar artery occlusion (proximal, middle, distal part), and further matched by the National Institutes of Health Stroke Scale score on admission to hospital (0-4, 4-15,16-20, 21-42), premorbid Modified Rankin Scale score, MSCT brain findings on admission to hospital (ischemia/ no ischemia), time from symptom onset to treatment (0-3h, 3-6h, later than 6 h), age (+/- 5 years), type of treatment (conservative treatment, intravenous thrombolysis with alteplase, mechanical thrombectomy, intravenous thrombolysis with alteplase + mechanical thrombectomy), type of mechanical thrombectomy (intracranial basilar artery stenting performed/not performed), and comorbid arterial hypertension (yes or no).

The data for historical controls will be obtained retrospectively from the Central Hospital Database which contains demographic, clinical, laboratory, and neuroimaging records of all patients with posterior circulation stroke secondary to basilar artery occlusion treated in the same Center from January 2015 to May 2024. The data will be analyzed, and the results will be compared between the investigational group and historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute basilar artery occlusion confirmed on MSCT/ MR angiography
* Premorbid mRS ≤ 3
* Signed written consent

Exclusion Criteria:

* Hypersensitivity to one of the components of the drug
* Breastfeeding and pregnancy
* Epilepsy, epileptic seizure
* Severe renal impairment (grade IV and V)
* Ischemic stroke in the previous three months
* Metastatic cancer
* Sepsis or a severe infection on admission
* Acute coronary syndrome, pulmonary embolism, and deep venous thrombosis on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants in the Cerebrolysin group with the Modified Rankin Scale (mRS) score 0-3 at 90 days post-stroke compared to historical controls | 90 days (3 months) after the stroke
  The functional outcomes will be assessed using the Modified Rankin Scale (mRS), with scores ranging from 0 (best functional outcome) to 6 (worst functional outcome). In the context of posterior circulation stroke, a favorable functional outcome is defined as an mRS score of ≤3 on day 90 post-stroke.
Mortality rate in the Cerebrolysin group compared to historical controls | 90 days (3 months) after the stroke
  The mortality rate will be assessed using the Modified Rankin Scale, which ranges from 0 to 6, where a score of 6 corresponds to the "death" outcome.

SECONDARY OUTCOMES:
Change in any and symptomatic intracerebral bleeding in the Cerebrolysin group compared to historical controls | 24 hours and 14 days after the stroke
  The follow-up computed tomography scans will be performed 24 hours and 14 days after the stroke. Additional scans will be obtained when indicated (before introducing anticoagulant therapy, in case of clinical deterioration with an increase of ≥4 points on the NIHSS from baseline or the lowest value within 7 days, in case of death, or for other reasons).
  Types of intracerebral bleeding and symptomatic intracerebral bleeding will be classified according to the ECASS III trial classification. Other types of bleeding which cannot be classified by ECASS III classification will be listed as "other".
Change in the National Institutes of Health Stroke Scale (NIHSS) compared to historical controls | 24 hours, 14 days, and 90 days after the stroke
  The clinical outcomes will be evaluated using the National Institutes of Health Stroke Scale (NIHSS), which ranges from 0 to 42. Lower scores indicate a better clinical outcome, while higher scores indicate a worse outcome.
  A change of at least 2 points on the National Institutes of Health Stroke Scale (NIHSS) is considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Roje Bedeković, MD, PhD, Principal Investigator — Sestre milosrdnice University Hospital Center

REFERENCES:
- [Background] Hawkes MA, Blaginykh E, Ruff MW, Burrus T, Wijdicks EFM, Rabinstein AA. Long-term mortality, disability and stroke recurrence in patients with basilar artery occlusion. Eur J Neurol. 2020 Mar;27(3):579-585. doi: 10.1111/ene.14126. Epub 2019 Dec 8. PMID 31721389
- [Background] Smith WS, Lev MH, English JD, Camargo EC, Chou M, Johnston SC, Gonzalez G, Schaefer PW, Dillon WP, Koroshetz WJ, Furie KL. Significance of large vessel intracranial occlusion causing acute ischemic stroke and TIA. Stroke. 2009 Dec;40(12):3834-40. doi: 10.1161/STROKEAHA.109.561787. Epub 2009 Oct 15. PMID 19834014
- [Background] Lang W, Stadler CH, Poljakovic Z, Fleet D; Lyse Study Group. A prospective, randomized, placebo-controlled, double-blind trial about safety and efficacy of combined treatment with alteplase (rt-PA) and Cerebrolysin in acute ischaemic hemispheric stroke. Int J Stroke. 2013 Feb;8(2):95-104. doi: 10.1111/j.1747-4949.2012.00901.x. Epub 2012 Sep 26. PMID 23009193
- [Background] Khasanova DR, Kalinin MN. Cerebrolysin as an Early Add-on to Reperfusion Therapy: Risk of Hemorrhagic Transformation after Ischemic Stroke (CEREHETIS), a prospective, randomized, multicenter pilot study. BMC Neurol. 2023 Mar 27;23(1):121. doi: 10.1186/s12883-023-03159-w. PMID 36973684
- [Background] Guekht A, Vester J, Heiss WD, Gusev E, Hoemberg V, Rahlfs VW, Bajenaru O, Popescu BO, Doppler E, Winter S, Moessler H, Muresanu D. Safety and efficacy of Cerebrolysin in motor function recovery after stroke: a meta-analysis of the CARS trials. Neurol Sci. 2017 Oct;38(10):1761-1769. doi: 10.1007/s10072-017-3037-z. Epub 2017 Jul 13. PMID 28707130
- [Background] Poljakovic Z, Supe S, Ljevak J, Starcevic K, Peric I, Blazevic N, Krbot-Skoric M, Jovanovic I, Ozretic D. Efficacy and safety of Cerebrolysin after futile recanalisation therapy in patients with severe stroke. Clin Neurol Neurosurg. 2021 Aug;207:106767. doi: 10.1016/j.clineuro.2021.106767. Epub 2021 Jun 18. PMID 34214867
- [Background] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396